CLINICAL TRIAL: NCT01150084
Title: "Step by Step": A Feasibility Study of the Promotion of Lunchtime Walking to Increase Physical Activity and Improve Mental Well-being in Sedentary Employees
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Collaborators: BUPA Foundation (Other)
Responsible Party: Dr Cecilie Thogersen-Ntoumani, University of Birmingham
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: ISRCTN01150084; ISRCTN01150084 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2009-09

CONDITIONS: Exercise; Sedentary
Keywords: increasing physical activity in sedentary employees
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Treatment Delay

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lunchtime walking (Experimental)
  Interventions: Other: 16-week lunchtime walking intervention
- waiting-list control (Other)
  Interventions: Other: delayed treatment

INTERVENTIONS:
Other: 16-week lunchtime walking intervention — 10 week group led lunchtime walks (each 30 minutes) followed by 6 weeks independent walking
  Arms: lunchtime walking
Other: delayed treatment — to start at week 10
  Arms: waiting-list control

SUMMARY:
Increasing rates of sedentary living, often complemented by obesity, among large segments of the adult population are associated with costs to individual health and well-being and thereby to society as a whole. Although some workplaces offer physical activity opportunities, those employees who tend to need it the most (i.e., the health needy) are often not attracted. In this project, the investigators propose to develop and evaluate a programme that is targeted to the sedentary health needy employees. The investigators will work with the corporate partner (a large university) to attract such employees through an extensive social marketing driven campaign. A 16-week lunchtime walking programme is proposed in which walking groups are offered followed by support and motivational strategies for longer term independent walking. The investigators will examine the effects of the programme on total amount of walking (including a follow-up assessment 4 months later) and will use innovative technology (Smartphones) to also examine the effect of lunchtime walks on well-being and work performance within and between participants.

ELIGIBILITY:
Inclusion Criteria:

* healthy, mobile, 18-65 year old employees who report they are engaging in less than 30 minutes of moderate intensity physical activity per week

Exclusion Criteria:

* employees with significant auditory or visual problems and those who have severe musculoskeletal disorders that prevent them from engaging in physical activity. Medical clearance will be requested for those who report any cardiovascular disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
number of steps | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie Thogersen-Ntoumani, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, West Midlands, United Kingdom